CLINICAL TRIAL: NCT02147574
Title: Laparoscope Subtotal Colectomy With Anti-peristaltic Ileo-sigmoid Anastomosis for the Treatment of Slow-transit Constipation:Therapeutic Evaluation
Brief Title: Anti-peristaltic Ileo-sigmoid Anastomosis for the Treatment of Slow-transit Constipation:Therapeutic Evaluation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anlong Zhu (Other)
Responsible Party: Sponsor-Investigator, Anlong Zhu, Vice Chairman, First Affiliated Hospital of Harbin Medical University
Organization: First Affiliated Hospital of Harbin Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: zhuanlone0001; fahhmuzal0001 (Other: FirstAHHarbinMU)
Record Dates: First submitted 2014-05-08; First posted 2014-05-28 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Constipation
Keywords: slow-transit constipation; laparoscope Sub-total Colectomy; anti-peristaltic anastomosis
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- antiperistaltic ileosigmoid anastomosis (Experimental): To assess the operative results after laparoscope subtotal colectomy with antiperistaltic ileosigmoid anastomosis for the slow-transit constipation.
  Interventions: Procedure: Anti-peristaltic ileosigmoid anastomosis

INTERVENTIONS:
Procedure: Anti-peristaltic ileosigmoid anastomosis — 1,Laparoscope Sub-total Colectomy： After the entire colon mobilization,the ileum is resected at 10cm from ileocecum and 10-15cm colon up to peritoneal reflection is reserved. The ileocolic artery should be reserved carefully.2, Intestinal tract reconstruction: The terminal ileum is turned over 180°in anti-clockwise direction along the superior mesenteric vein long axis. To avoid the small mesenteric torsion , we should turn the broken edge towards inside. The terminal ileum and 10-15cm colon anastomose in anti-peristaltic direction,the anastomotic length is 8-10 cm.3, Sewn the space between anastomotic Intestine and posterior peritoneum. A drain is placed in the abdominal cavity and another one is placed in anal canal.

SUMMARY:
Purpose:

To evaluate the curative effect of Laparoscope Sub-total Colectomy with Anti-peristaltic ileosigmoid anastomosis for the treatment of slow-transit constipation on the patients with STC.

Methods and techniques:

The data of patients with STC preformed surgery of laparoscopic subtotal colectomy with anti-peristaltic ileosigmoid anastomosis during 2009.01-2014.05 was reviewed. The related status such as frequency of defecation, course of constipation, laxatives use condition the condition of using laxatives, and changes in weight were investigated. Changes of defecation and weight, periprocedural complications (wound infection, lung infection and intestinal fistula), long-term complication (malnutrition, abdominal pain, ileus), life satisfaction, wexner score of pre-operation and postoperation ect were investigated in follow-ups.

DETAILED DESCRIPTION:
Theoretical Basis:

As far as the current research status, total colectomy or subtotal colectomy has become the preferred type of surgery for slow-transit constipation treatment. There are different opinions on intestinal anastomosis and the specific scope of excision. There is a type of surgery reserving the ileocecum, as the ileocaecal valve has the function of postponing the fecal evacuation. There's also a type of surgery excising the ileocecum , and establishing the pouch, as reserving the ileocecum may cause the recurrence of constipation, and establishing the pouch has function of relieving the postoperative fecal incontinence. On the basis, our own type of surgery is designed; ileocecum is excised for preventing the recurrence of constipation, while the anti-peristaltic ileosigmoid anastomosis between the small intestine and part of sigmoid is made for preventing the severe diarrhea.

Methods and techniques:

The data of patients with STC preformed surgery of laparoscopic subtotal colectomy with anti-peristaltic ileosigmoid anastomosis during 2009.01-2014.05 was reviewed. The related status such as frequency of defecation, course of constipation, laxatives use condition the condition of using laxatives, and changes in weight were investigated. Changes of defecation and weight, periprocedural complications (wound infection, lung infection and intestinal fistula), long-term complication (malnutrition, abdominal pain, ileus), life satisfaction, wexner score of pre-operation and postoperation ect were investigated in follow-ups.

Surgical operation process:

1,Laparoscope Sub-total Colectomy： After the entire colon mobilization,the ileum is resected at 10cm from ileocecum and 10-15cm colon up to peritoneal reflection is reserved. The ileocolic artery should be reserved carefully.2, Intestinal tract reconstruction: The terminal ileum is turned over 180°in anti-clockwise direction along the superior mesenteric vein long axis. To avoid the small mesenteric torsion, we should turn the broken edge towards inside. The terminal ileum and 10-15cm colon anastomose in anti-peristaltic direction,the anastomotic length is 8-10 cm.3, Sewn the space between anastomotic Intestine and posterior peritoneum. A drain is placed in the abdominal cavity and another one is placed in anal canal.

ELIGIBILITY:
Inclusion Criteria:

* the clinical diagnose of STC
* Severe symptoms of constipation, defecating less than 2 times per week, no awareness of defecation, using laxatives to help defecation or there's no effects of laxatives.
* Symptoms of constipation last at least 2 years, and ineffective effects received from medicine treatment for more than one year.
* Colorectal organic disease was excluded
* More than one colonic transit trials suggest dysfunction of colon transport, no significant intestinal transit dysfunction

Exclusion Criteria:

* significant mental disorder
* surgical contraindications
* Can't accept surgery subjectively

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-12; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Improvement of signs and symptoms associated with constipation complication | preoperative, and at 6 months postoperative

SECONDARY OUTCOMES:
Improvement of signs and symptoms associated with constipation complication | preoperative, at 12 months postoperative

CONTACTS AND LOCATIONS:
Overall Officials: anlong zhu, postdoctor, Study Chair — First Affiliated Hospital of Harbin Medical University
Locations (1):
- The First Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang, China